CLINICAL TRIAL: NCT06673056
Title: Effects of N-Acetyl-L-Leucine on Ataxia-Telangiectasia (A-T: A Phase III, Randomized, Placebo-controlled, Double-blind, Crossover Study
Brief Title: A Pivotal Study of N-Acetyl-L-Leucine on Ataxia-Telangiectasia (A-T)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IntraBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IB1001-303
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Ataxia-Telangiectasia; Ataxia-Telangiectasia (A-T)
Keywords: Ataxia-Telangiectasia; Louis Bar Syndrome
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — acetylleucine; IB1001

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, crossover, multi-center, study with 1:1 randomization of IB1001 plus SOC for 12-weeks versus placebo plus SOC for 12-weeks, followed by open-label extension study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetyl-L-leucine (IB1001) (Experimental): Oral administration (granule in a sachet for suspension in water, orange juice, or almond milk). Patients will receive a total daily dose of 2-4 g/day based on weight-tiered doses.
  Interventions: Drug: N-Acetyl-L-Leucine
- Placebo comparator (Placebo Comparator): Oral administration (granule in a sachet for suspension in water, orange juice, or almond milk). Patients will receive a total daily dose of 2-4 g/day based on weight-tiered doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-Acetyl-L-Leucine — N-Acetyl-L-Leucine is a modified amino-acid ester that is orally administered (granules for suspension in a sachet)
  Other Names: IB1001; levacetylleucine
  Arms: N-acetyl-L-leucine (IB1001)
Other: Placebo — Matching Placebo Sachet
  Arms: Placebo comparator

SUMMARY:
A pivotal, randomized, double-blind, placebo-controlled, multi-center therapeutic study for patients age 4 and older with a confirmed diagnosis of Ataxia-Telangiectasia (A-T). The objective of this study is to evaluate the safety, tolerability and efficacy of N-acetyl-L-leucine (IB1001) compared to standard of care.

DETAILED DESCRIPTION:
This is a multinational, randomized, placebo-controlled, double-blinded, cross-over Phase III study that will assess the safety and efficacy of N-Acetyl-L-Leucine (IB1001) versus Placebo for the treatment of Ataxia-Telangiectasia (A-T).

Patients will be assessed during three study periods: a baseline period (approximately 2-weeks), after which they will be randomized (1:1) to receive treatment with IB1001 or Placebo for approximately 12-weeks during the first intervention period ("Period I"). Following Period I, patients will crossover to receive the opposite treatment (IB1001 or Placebo) for approximately 12-weeks during a second intervention period ("Period II).

Patients will be assessed twice during each study period. Patients who have participated in the study may be offered the opportunity to roll over into an Extension Phase, which is planned to allow patients to have further access to IB1001.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent signed by the patient and/or their legal representative / parent/ impartial witness 2. Male or female aged ≥4 years with a genetically confirmed diagnosis of A-T at the time of signing informed consent.

  3. Females of childbearing potential, defined as a premenopausal female capable of becoming pregnant, will be included if they are either sexually inactive (sexually abstinent for 14 days prior to the first dose and confirm to continue through 28 days after the last dose) or using one of the following highly effective contraceptives (i.e. results in <1% failure rate when used consistently and correctly) 14 days prior to the first dose continuing through 28 days after the last dose:
  1. intrauterine device (IUD);
  2. surgical sterilization of the partner (vasectomy for 6 months minimum);
  3. combined (estrogen or progestogen containing) hormonal contraception associated with the inhibition of ovulation (either oral, intravaginal, or transdermal);
  4. progestogen only hormonal contraception associated with the inhibition of ovulation (either oral, injectable, or implantable);
  5. intrauterine hormone releasing system (IUS);
  6. bilateral tubal occlusion. 4. Females of non-childbearing potential who have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

  <!-- -->

  1. hysteroscopic sterilization;
  2. bilateral salpingectomy;
  3. hysterectomy;
  4. bilateral oophorectomy; OR be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status. FSH analysis for postmenopausal women will be done at screening. FSH levels should be in the postmenopausal range as determined by the central laboratory.

     5. Non-vasectomized male patient agrees to use a condom with spermicide during the study until 90 days beyond the last dose of study medication and the female partner agrees to comply with inclusion criteria 3 or 4. For a vasectomized male who has had his vasectomy 6 months or more prior to study start, it is required that they use a condom during sexual intercourse. A male who has been vasectomized less than 6 months prior to study start must follow the same restrictions as a non-vasectomized male.

     6. If male, patient agrees not to donate sperm from the first dose until 90 days after their last dose.

     7. Patients must fall within:

  <!-- -->

  1. A SARA score of 7 ≤ X ≤ 34 points (out of 40) AND
  2. Either:

  i. Within the 2-7 range (0-8 range) of the Gait subtest of the SARA scale OR ii. Be able to perform the 9-Hole Peg Test with Dominant Hand (9HPT-D) (SCAFI subtest) in 20 ≤ X ≤150 seconds.

  8. Weight ≥15 kg at screening. 9. Patients are willing to disclose their existing medications/therapies for (the symptoms) of A-T, including those on the prohibited medication list. Non-prohibited medications/therapies, therapy, and physiotherapy) are permitted provided:
  1. The Investigator does not believe the medication/therapy will interfere with the study protocol/results
  2. Patients have been on a stable dose/duration and type of therapy for at least 42 days before Visit 1 (Baseline 1)
  3. Patients are willing to maintain a stable dose/do not change their therapy throughout the duration of the study.

     10. An understanding of the implications of study participation, provided in the written patient information and informed consent by patients or their legal representative/parent, and demonstrates a willingness to comply with instructions and attend required study visits (for children this criterion will also be assessed in parents or appointed guardians).

     Exclusion Criteria:
* 1. Patients who have any known hypersensitivity or history of hypersensitivity to:

  1. Acetyl-Leucine (DL-, L-, D-) or derivatives.
  2. Excipients the IB1001 sachet (namely isomalt, hypromellose, and strawberry flavor).
  3. Excipients the placebo sachet (namely isomalt, hypromellose, strawberry flavor, citric acid, microcrystalline cellulose, lactose, denatonium benzoate).

     2. Simultaneous participation in another clinical study or participation in any clinical study involving administration of an investigational medicinal product (IMP; 'study drug') for at least 42 days prior to Visit 1. At the discretion of the investigator, Medical Monitor, and Sponsor, the washout period for specific IMPs may be longer based on the pharmacological activity and pharmacokinetics of the drug.

     3. Patients with a physical or psychiatric condition which, at the investigator's discretion and in consultation with the Medical Monitor and Sponsor (as applicable), may put the patient at risk, may confound the study results, or may interfere with the patient's participation in the clinical study, i.e. reliably perform study assessments.

     4. Known or persistent use, misuse, or dependency of medication, drugs, or alcohol.

     5. Current or planned pregnancy or women who are breastfeeding. 6. Patients with severe vision or hearing impairment (that is not corrected by glasses or hearing aids) that, at the investigator's discretion, interferes with their ability to perform study assessments.

     7. Patients who have been diagnosed with arthritis or other musculoskeletal disorders affecting joints, muscles, ligaments, and/or nerves that by themselves affects patient's mobility and, at the investigator's discretion, interferes with their ability to perform study assessments.

     8. Patients unwilling and/or not able to undergo a 42-day washout period from any of the following prohibited medication prior to Visit 1 (Baseline 1) and remain without prohibited medication through Visit 6.

  <!-- -->

  1. N-Acetyl-DL-Leucine (e.g. Tanganil®);
  2. N-Acetyl-L-Leucine (prohibited if not provided as IMP in the IB1001-303 trial);
  3. Sulfasalazine;
  4. Rosuvastatin.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia | End of Period I (week 12) vs. End of Period 2 (week 24)
  The Scale for Assessment and Rating of Ataxia has 8 items that are related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements, and heel-shin test. The range is 0-40 points, with a lower score representing neurological improvement and a higher score representing neurological worsening.

SECONDARY OUTCOMES:
Spinocerebellar Ataxia Functional Index (SCAFI) | End of Period I (week 12) vs. End of Period 2 (week 24)
  Spinocerebellar Ataxia Functional Index (SCAFI) is composed of 8 Meter Walk Test, 9-Hole Peg Test of Dominant and Non-Dominant Hand (9HPT-D/9HPT-ND) (the 3 tests are timed assessments; each is done twice and values are averaged; the 8MWT and 9HPT-D and 9HPT-ND values are converted from times to rates, and the results expressed as a composite Z-score of each test relative to baseline) and the PATA rate (counted number how often a patient can repeat the syllables "PATA" within 10 seconds), a measure of speech performance. The scores of these 3 were transformed to Z-scores (=individual's average of both trials to perform the respective task - mean of study population at baseline) / SD of study population at baseline). A Z-score of 0 equates to the population mean at baseline. For all 3, higher Z-scores (above mean) mean better performance. The SCAFI total score was calculated as the arithmetic mean of the non-missing Z-scores for the 3. A higher total score means better performance.
Physician's / Caregiver's / Patient's Clinical Global Impressions (CGI) | End of Period I (week 12) vs. End of Period 2 (week 24)
  The Clinical Global Impression of Improvement assessed by the investigator/caregiver/patient is evaluated on a 7 point Likert scale ranging from 1='very much improved' to 7='very much worse'
EuroQuol- 5 Dimension (EQ-5D) Quality of Life Scale | End of Period I (week 12) vs. End of Period 2 (week 24)
  For posting, health-related quality of life based on the EQ-5D visual analogue scale (VAS) was presented as a secondary endpoint.
  EQ-5D VAS is a 0-100 scale where patients are asked to indicate their overall health, with a score of 0 indicating worst health and a score of 100 indicating best health.
International Cooperate Ataxia Rating Scale (ICARS) | End of Period I (week 12) vs. End of Period 2 (week 24)
  The International Cooperate Ataxia Rating Scale (ICARS) was developed to quantify the level of impairment as a result of ataxia as related to hereditary ataxias. Disorders rated as subscales within the ICARS are: Postural and gait disturbances, Limb Ataxia, Dysarthria, and Oculomotor disorders
Neuro Quality of Life - Upper Extremity Function (NeuroQOL-UEF) | End of Period I (week 12) vs. End of Period 2 (week 24)
  The Neurology Quality of Life (NeuroQOL) Upper Extremity Function (UEF) scale is a self-report of health-related quality of life that measures the patient's ability to carry out various activities involving digital, manual, and reach-related functions, ranging from fine motor to self-care (activities of daily living)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - The University of Texas Health (UT Health), Houston, Texas
- Germany (2):
  - University of Cologne, Cologne
  - University of Giessen, Giessen
- Slovakia (2):
  - Comenius University Bratislava, Bratislava
  - University Hospital L. Pasteur, Košice
- Hospital Universitario La Paz, Madrid, Spain
- University of Bern, Bern, Switzerland
- United Kingdom (2):
  - Royal Papworth Hospital, Cambridge
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published within a reasonable timeframe of completion. Pseudonymised individual patient data may be available in these findings.